CLINICAL TRIAL: NCT04249674
Title: Impact of CYP2D6 Genetic Polymorphism on the Vulnerability to Drug-drug Interactions With Tramadol: a Gene-environment Interaction and Phenoconversion Study on Patients Undergoing a Steady Treatment With a Potent CYP2D6 Inhibitor.
Brief Title: Impact of CYP2D6 Genetic Polymorphisms on the Vulnerability to Drug-drug Interactions With Tramadol
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Youssef Daali (Unknown); Jules Desmeules (Unknown); Kenza Abouir (Unknown); Eduardo Schiffer (Unknown); Bernard Walder (Unknown)
Responsible Party: Principal Investigator, Caroline Samer, Doctor, University Hospital, Geneva
Other Study IDs: 2019-01418
Record Dates: First submitted 2019-12-04; First posted 2020-01-31 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Interaction; Pain
Keywords: Cytochrome; Polymorphism; Genotyping; Phenotyping; Tramadol; CYP2D6 inhibitor; Phenoconversion; Environment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological fluids : blood, urine and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient under a CYP2D6 inhibitor and under Tramadol
  Interventions: Diagnostic Test: Dextrometorphan; Genetic: Genotyping by single nulcetoide polymorphism.
- Patient not under a CYP2D6 inhibitor but under Tramadol
  Interventions: Diagnostic Test: Dextrometorphan; Genetic: Genotyping by single nulcetoide polymorphism.

INTERVENTIONS:
Diagnostic Test: Dextrometorphan — Administration of 4 ml=10 mg of Dextrometorphan (Bexine sirup)
Genetic: Genotyping by single nulcetoide polymorphism. — Single nucleotide polymorphism determination

SUMMARY:
Despite its poor abundance in the liver, CYP2D6 is the second most important CYP in drug metabolism, metabolizing 20% of drugs. The high inter-individual variability in CYP2D6 expression is explained by genetic variations, but also by drug-drug interactions (DDIs). Recent studies have pointed out the poor therapeutic predictable value of DDI. Indeed, the clinical outcomes of a DDI may involve several intrinsic factors affecting the vulnerability to and extent of DDI, such as genetic polymorphisms, comorbidities, age and sex.

In this regard, the present research project aims to investigate the effect of genetic polymorphism on DDIs involving CYP2D6 (gene-environment interaction) and its implications for tramadol efficacy and safety in a clinical setting. In a previous study, we demonstrated differences in both the rate of phenoconversion and the magnitude of DDI in healthy volunteers, that were either heterozygote normal metabolizers (NMs) carrying a non-functional CYP2D6 allele (activity score (AS) 1) and homozygous NM carrying two fully-functional CYP2D6 alleles (AS 2).

This prospective study will include patients scheduled for a general surgery of less than 3 hours and planned to be treated with oral tramadol as a routine post-operative pain management.

Patients taking part in the study may receive diagnosis, therapeutic or other interventions but the groups of individuals (controls vs inhibited) are predefined based on the routine treatment of the patients.

There will be no assigned specific interventions to the study participants and CYP2D6 phenotypes will be classified in five activity score groups (0.5, 1, 1.5, 2, >2) in the absence or presence of a potent CYP2D6 inhibitor received as part of routine medical care.

PK of tramadol and its active metabolite (M1), as well as its analgesic and PD effects and safety, will be compared between groups. Finally, the data generated will be used to build a physiologically-based PK (PBPK) model for tramadol in different sub-groups. The model will aim to predict the effect of CYP2D6 inhibition in virtual populations with different genetically-related CYP2D6 activities. This should allow prospective dose adjustment of tramadol (or appropriate drug selection) based on patients' genotype in the presence of a CYP2D6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Any male and female patients > 18 years scheduled for a surgery of less than 3 hours duration and planned to be treated with oral tramadol as a routine management of post-operative pain;
* Patients with physical conditions classified as ASA I to III, based on American Society of Anesthesiology classification;
* Patients treated chronically with a potent CYP2D6 inhibitor (for CYP2D6-inhibited arms only);
* Understanding of French language and able to give a written inform consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Any pathologies, use of drugs or food that may affect CYP activity (for control arms only and based on the 'drug interactions and cytochromes P450' table published by The Service of clinical Pharmacology and Toxicology [3], HUG and on the investigator's knowledge)
* Liver transplantation history
* Sensitivity to dextromethorphan (CYP2D6 probe drug) or any contra-indication to dextrometorphan
* Medical history of cirrhosis (Child Pugh B and C) or/and hepatosteatosis.
* Glomerular filtration rate (GFR) < 30 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through a pre-surgery anesthetic evaluation visit. During their scheduled visit with an anaesthesiologist, potential patients will be invited to participate to an information session where project aim and design, procedures involved, expected duration as well as possible risks will be explained in details.
  After sufficient time of reflection, volunteers willing to participate in the study will sign the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assess the proportion of patients in each group who acquires a phenotype switch (phenoconversion) with or without CYP2D6 inhibitor. | 10 hours

SECONDARY OUTCOMES:
Comparison of Tramadol , Dexrometorphan and their metabolites maximum plasma concentration (Cmax) according to patient belonging to the control or inhibited group. | 24 hours
Comparison of Tramadol, Dextrometorphan and their metabolites Area Under the curve (AUC) according to patient belonging to the control or to the inhibited group and to his CYP2D6 phenotype | 24 hours
Comparison of Tramadol, Dextrometorphan and their metabolites Clearance (CL) according to patient belonging to the control or to the inhibited group. | 24 hours

OTHER OUTCOMES:
Urinary metabolic ratio (UMR) tramadol/M1 in urine collection | 8 hours
Saliva metabolic ratio tramadol/M1 | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Daali, Pr., Study Director — University Hospital, Geneva; Caroline Samer, Doctor, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, HUG, Geneva, Switzerland